CLINICAL TRIAL: NCT06210295
Title: What is Behind Anemia in Systemic Lupus Erythematosus With Special Reference to Referactory Anemia
Brief Title: Anemia in Systemic Lupus Erythematosus Specially Refractory Type
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shymaa Saber, What is behind anemia in systemic lupus erythematosus with special reference to refractory anemia, Assiut University
Other Study IDs: 121293
Record Dates: First submitted 2023-12-13; First posted 2024-01-18 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Refractory Anemia in Systemic Lupus Erythematosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Anemia and Systemic lupus erythematosus: Systemic lupus patients with anemia and searching for causes of anemia and what is the most common and what are the causes of refractory anemia and relation of bone marrow affection
  Interventions: Combination Product: Laboratory investigtions

INTERVENTIONS:
Combination Product: Laboratory investigtions — To study causes of anemia in SLE in our environment and causes of refractory type and its relation to bone marrow affection and different drugs used in SLE
  Other Names: Bone marrow study

SUMMARY:
Systemic lupus erythroematosis (SLE) is a systemic autoimmune disease with multisystemic involvement. The condition has several phenotypes, with varying clinical presentations from mild mucocutaneous manifestations to multiorgan and severe central nervous system involvement. Several immunopathogenic pathways play a role in the development of SLE. Despite recent advances in technology and understanding of the pathological basis and risk factors for SLE, the exact pathogenesis is still not well known. Diagnosis of SLE can be challenging, and while several classification criteria have been posed, their utility in the clinical setting is still a matter of debate. Management of SLE is dictated by organ system involvement. Despite several agents shown to be efficacious in treating SLE, the disease still poses significant morbidity and mortality risks in patients[1].

Haematological abnormalities are common in systemic lupus erythroematosis. Anemia is found in about 50% of patients.

DETAILED DESCRIPTION:
Causes of anemia in SLE:

Anemia due to chronic disease is the most frequent in patients with SLE, representing approximately one-third of the cases [2].

Iron deficiency anemia is also a common cause, usually caused by blood loss (menorrhagia or gastrointestinal bleeding) [3].

Autoimmune hemolytic anemia (AIHA) a classification criteria for SLE [4]. The mechanism is thought to be caused by the destruction of red blood cells through warm or cold antibodies [5]. Patients with AIHA may present with symptoms of anemia or hemolysis or symptoms of an underlying disorder. Severe hemolysis may lead to hepatosplenomegaly, hemoglobinuria, and signs of heart failure [6]. Maanaging patients with AIHA may be challenging because specific therapy should be individualized in accordance with the disease manifestations and its severity [7].

Hemopoietic failure is the suspected to be the result of an immunologically damaged bone marrow (BM) .

Overall, hypocellularity, morphological dysplasia, increased fibrosis, and BM necrosis were common findings in patients with SLE with hemocytopenias, suggesting a primary BM involvement in pathogenesis of the disease, probably mediated by auto-antibodies, immune complexes, and immunopotent T cells [8, 9].

Solid proof of the participation of humoral immune mechanisms in hemopoietic dysfunction was obtained from patients with SLE with aplastic anemia, a BM failure syndrome of a definite immune pathogenesis [10-12].

In these cases, complement dependent or independent autoantibodies were found to suppress erythroid and granulocytic colony formation of BM progenitor cells [10-12].

Targeted by autoantibodies, the progenitor BM cells lead to various syndromes of hemopoietic failure, such as aplastic anaemia, hypoplasia of myeloid line, amegakaryocytic thrombocytopenia, and the extremely rare pure red cell aplasia (PRCA) [13-19].

The presence of the inhibitory autoantibody is typically related to SLE activity and can be suppressed by successful treatment-that is, by immunosuppression. However, PRCA can occur in the absence of disease activity or even precede the appearance of SLE [15].

In our study we will search for the most common causes of anemia in SLE in our environment ,focusing on the most common causes of refractory anemia in SLE.

ELIGIBILITY:
Inclusion Criteria:

* -Adult patients (≥18 years) satisfying 2019 EULAR/ACR classification for systemic lupus erythroematosis[24].
* Patients satisfying WHO criteria definition of anemia.

Exclusion Criteria:

* Mixed connective tissue disorders.
* Pregnancy .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient diagnosed as systemic lupus erythematosus with anemia aged more than 18 year old
Sampling Method: Probability Sample
Enrollment: 67 (Estimated)
Dates: Start 2024-07-09 (Estimated); Primary Completion 2024-09-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Causes of anemia | One week
  Assess causes of anemia in SLE and which of them is most common in our locality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Molina-Rios S, Rojas-Martinez R, Estevez-Ramirez GM, Medina YF. Systemic lupus erythematosus and antiphospholipid syndrome after COVID-19 vaccination. A case report. Mod Rheumatol Case Rep. 2023 Jan 3;7(1):43-46. doi: 10.1093/mrcr/rxac018. PMID 35246682
- [Background] Voulgarelis M, Kokori SI, Ioannidis JP, Tzioufas AG, Kyriaki D, Moutsopoulos HM. Anaemia in systemic lupus erythematosus: aetiological profile and the role of erythropoietin. Ann Rheum Dis. 2000 Mar;59(3):217-22. doi: 10.1136/ard.59.3.217. PMID 10700431
- [Background] Levine AB, Erkan D. Clinical assessment and management of cytopenias in lupus patients. Curr Rheumatol Rep. 2011 Aug;13(4):291-9. doi: 10.1007/s11926-011-0179-5. PMID 21503695
- [Background] Aringer M, Costenbader K, Daikh D, Brinks R, Mosca M, Ramsey-Goldman R, Smolen JS, Wofsy D, Boumpas DT, Kamen DL, Jayne D, Cervera R, Costedoat-Chalumeau N, Diamond B, Gladman DD, Hahn B, Hiepe F, Jacobsen S, Khanna D, Lerstrom K, Massarotti E, McCune J, Ruiz-Irastorza G, Sanchez-Guerrero J, Schneider M, Urowitz M, Bertsias G, Hoyer BF, Leuchten N, Tani C, Tedeschi SK, Touma Z, Schmajuk G, Anic B, Assan F, Chan TM, Clarke AE, Crow MK, Czirjak L, Doria A, Graninger W, Halda-Kiss B, Hasni S, Izmirly PM, Jung M, Kumanovics G, Mariette X, Padjen I, Pego-Reigosa JM, Romero-Diaz J, Rua-Figueroa Fernandez I, Seror R, Stummvoll GH, Tanaka Y, Tektonidou MG, Vasconcelos C, Vital EM, Wallace DJ, Yavuz S, Meroni PL, Fritzler MJ, Naden R, Dorner T, Johnson SR. 2019 European League Against Rheumatism/American College of Rheumatology Classification Criteria for Systemic Lupus Erythematosus. Arthritis Rheumatol. 2019 Sep;71(9):1400-1412. doi: 10.1002/art.40930. Epub 2019 Aug 6. PMID 31385462
- [Background] Jager U, Barcellini W, Broome CM, Gertz MA, Hill A, Hill QA, Jilma B, Kuter DJ, Michel M, Montillo M, Roth A, Zeerleder SS, Berentsen S. Diagnosis and treatment of autoimmune hemolytic anemia in adults: Recommendations from the First International Consensus Meeting. Blood Rev. 2020 May;41:100648. doi: 10.1016/j.blre.2019.100648. Epub 2019 Dec 5. PMID 31839434
- [Background] Hill QA, Stamps R, Massey E, Grainger JD, Provan D, Hill A; British Society for Haematology. The diagnosis and management of primary autoimmune haemolytic anaemia. Br J Haematol. 2017 Feb;176(3):395-411. doi: 10.1111/bjh.14478. Epub 2016 Dec 22. No abstract available. PMID 28005293
- [Background] Trindade VC, Carneiro-Sampaio M, Bonfa E, Silva CA. An Update on the Management of Childhood-Onset Systemic Lupus Erythematosus. Paediatr Drugs. 2021 Jul;23(4):331-347. doi: 10.1007/s40272-021-00457-z. Epub 2021 Jul 10. PMID 34244988
- [Background] Pereira RM, Velloso ER, Menezes Y, Gualandro S, Vassalo J, Yoshinari NH. Bone marrow findings in systemic lupus erythematosus patients with peripheral cytopenias. Clin Rheumatol. 1998;17(3):219-22. doi: 10.1007/BF01451051. PMID 9694056
- [Background] Feng CS, Ng MH, Szeto RS, Li EK. Bone marrow findings in lupus patients with pancytopenia. Pathology. 1991 Jan;23(1):5-7. doi: 10.3109/00313029109061430. PMID 2062568
- [Background] Bailey FA, Lilly M, Bertoli LF, Ball GV. An antibody that inhibits in vitro bone marrow proliferation in a patient with systemic lupus erythematosus and aplastic anemia. Arthritis Rheum. 1989 Jul;32(7):901-5. PMID 2751721
- [Background] Fitchen JJ, Cline MJ, Saxon A, Golde DW. Serum inhibitors of hematopoiesis in a patient with aplastic anemia and systemic lupus erythematosus. Recovery after exchange plasmapheresis. Am J Med. 1979 Mar;66(3):537-42. doi: 10.1016/0002-9343(79)91097-0. No abstract available. PMID 433958
- [Background] Brooks BJ Jr, Broxmeyer HE, Bryan CF, Leech SH. Serum inhibitor in systemic lupus erythematosus associated with aplastic anemia. Arch Intern Med. 1984 Jul;144(7):1474-7. PMID 6732407
- [Background] Kiely PD, McGuckin CP, Collins DA, Bevan DH, Marsh JC. Erythrocyte aplasia and systemic lupus erythematosus. Lupus. 1995 Oct;4(5):407-11. doi: 10.1177/096120339500400512. PMID 8563736
- [Background] Fisch P, Handgretinger R, Schaefer HE. Pure red cell aplasia. Br J Haematol. 2000 Dec;111(4):1010-22. doi: 10.1046/j.1365-2141.2000.02429.x. No abstract available. PMID 11167735
- [Background] Habib GS, Saliba WR, Froom P. Pure red cell aplasia and lupus. Semin Arthritis Rheum. 2002 Feb;31(4):279-83. doi: 10.1053/sarh.2002.30440. PMID 11836661
- [Background] Roffe C, Cahill MR, Samanta A, Bricknell S, Durrant ST. Aplastic anaemia in systemic lupus erythematosus: a cellular immune mechanism? Br J Rheumatol. 1991 Aug;30(4):301-4. doi: 10.1093/rheumatology/30.4.301. PMID 1863830
- [Background] Mavragani CP, Vlachaki E, Voulgarelis M. Pure red cell aplasia in a Sjogren's syndrome/lupus erythematosus overlap patient. Am J Hematol. 2003 Apr;72(4):259-62. doi: 10.1002/ajh.10302. PMID 12666137
- [Background] Charles RJ, Sabo KM, Kidd PG, Abkowitz JL. The pathophysiology of pure red cell aplasia: implications for therapy. Blood. 1996 Jun 1;87(11):4831-8. PMID 8639856
- [Background] Hartman KR, LaRussa VF, Rothwell SW, Atolagbe TO, Ward FT, Klipple G. Antibodies to myeloid precursor cells in autoimmune neutropenia. Blood. 1994 Jul 15;84(2):625-31. PMID 7517722
- [Background] Cappellini MD, Motta I. Anemia in Clinical Practice-Definition and Classification: Does Hemoglobin Change With Aging? Semin Hematol. 2015 Oct;52(4):261-9. doi: 10.1053/j.seminhematol.2015.07.006. Epub 2015 Jul 17. PMID 26404438
- [Background] Sonawale A, Pasiddhi S, Sabnis NH. Aetiology and outcome of anemia in patients with systemic lupus erythematosus. Int J Adv Med. 2017;4:968-73.
- [Background] Gladman DD, Ibanez D, Urowitz MB. Systemic lupus erythematosus disease activity index 2000. J Rheumatol. 2002 Feb;29(2):288-91. PMID 11838846